CLINICAL TRIAL: NCT07371338
Title: Dose-Escalation, Single-Center, Open-label Phase 1 Clinical Trial to Evaluate the Safety, Efficacy, and Pharmacokinetics of Adeno-associated Virus(AAV) Gene Therapy Product IPS101A in Parkinson's Disease Patients With Hoehn-Yahr Stage 4-5, Diagnosed in More Than 10 Years and Uncontrolled by All Available Monotherapy or Combination Therapy
Brief Title: Phase 1 Clinical Trial to Evaluate the Safety, Efficacy, and Pharmacokinetics of IPS101A in Parkinson's Disease Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innopeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPS101A-10
Record Dates: First submitted 2025-11-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease; Parkinson's Disease
Keywords: PD; AAV; Adeno-associated Virus; Gene therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose (1.0 x 10^10 vg/patient) (Experimental): IPS101A
  Interventions: Drug: IPS101A
- High dose(2.0 x 10^10 vg/patient) (Experimental): IPS101A
  Interventions: Drug: IPS101A

INTERVENTIONS:
Drug: IPS101A — The investigational product (IP) will be administered as a single dose. All subjects will receive stereotactic injections into the left and right substantia nigra of the midbrain, with one administration per side.

SUMMARY:
The purpose of this study is to evaluate the dose-related safety and tolerability of IPS101A, an adeno-associated virus (AAV) gene therapy, in patients with Parkinson's disease who exhibit severe functional impairment corresponding to Hoehn & Yahr stages 4-5 and whose symptoms are not adequately controlled despite all available monotherapy and combination therapy options. In addition, the study aims to assess the maximum tolerated dose (MTD) of IPS101A, as well as its preliminary efficacy and pharmacokinetic (PK) characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have a diagnosis of Parkinson's disease that meets the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria at the time of the Screening Visit.
2. Male or female subjects aged 50 to 80 years (inclusive) at the time of providing written informed consent, with a documented diagnosis of Parkinson's disease.
3. Subjects with a duration of Parkinson's disease of at least 10 years prior to the Screening Visit, based on medical history and/or medical records.
4. Subjects with Parkinson's disease that is inadequately controlled despite all available standard-of-care treatments, including monotherapy or combination therapy, as determined by the Investigator.
5. Subjects with a Hoehn & Yahr stage of 4 or 5 in the off state at the Screening Visit.

Exclusion Criteria:

1. Subjects with Parkinson's disease dementia (PDD) who meet the diagnostic criteria established by the Movement Disorder Society (MDS) Task Force, as determined by the Investigator at Screening.
2. Subjects with a Korean Mini-Mental State Examination (K-MMSE) score ≤ 24 at the Screening assessment.
3. Subjects in whom imaging findings suggestive of Parkinsonism-plus syndrome are observed on PET and MRI performed at the Screening Visit, as assessed by the Investigator and/or a qualified imaging specialist.
4. Subjects who do not meet the diagnostic criteria for Parkinson's disease dementia but present with major visual hallucinations, as judged by the Investigator.
5. Subjects with drug-induced parkinsonism, confirmed by clinical history and/or medical records, and determined by the Investigator.
6. Subjects who are judged by the investigator to be unsuitable for participation in this clinical trial.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation: dose-limiting toxicity (DLT) | Baseline to Week 8
  Frequency and proportion of subjects who developed dose-limiting toxicity (DLT)
Safety Evaluation: Severity and frequency of reported adverse events | Baseline to Week 52
  Assess severity and frequency of reported adverse events
Safety Evaluation: clinically-relevant changes in laboratory testing assessed by medical personnel | Baseline to Week 52
  The clinical significance of laboratory test results after administration of a clinical trial drug is confirmed by comparing them with those before administration.
Safety Evaluation: clinically-relevant changes in physical exams assessed by medical personnel | Baseline to Week 52
  The results of the physical examination after administration of the clinical trial drug are compared with those before administration to determine whether clinically significant symptoms occur.

SECONDARY OUTCOMES:
Change from Baseline in Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) scores (defined on/off) | Baseline to Weeks 4, 12, 24, 36, and 52.
  Each symptom is rated on a scale of 0 to 4, with higher scores indicating more severe Parkinson's disease.
Change from Baseline in Hoehn & Yahr stage (defined on/off) | Weeks 1, 4, 12, 24, 36, and 52.
  This scale is classified from 0 to 5, with a higher score indicating a more severe degree of Parkinson's disease.
Change from Baseline in Non-Motor Symptoms Scale for Parkinson's Disease (NMSS) | Weeks 4, 12, 24, 36, and 52.
  This scale is rated on a scale of severity (0-3 points) and frequency (1-4 points). A higher score indicates more severe Parkinson's disease.
Change from Baseline in Parkinson's Disease Questionnaire (PDQ-39) scores | Weeks 4, 12, 24, 36, and 52
  The scale consists of 800 points, and a higher score indicates a lower quality of life.
Distribution evaluation of IPS101A (AAV9 vector distribution evaluation)-CSF | Baseline to Week 52
  After IP administration, the detection of AAV genome was measured using q-PCR.
Distribution evaluation of IPS101A (AAV9 vector distribution evaluation)-blood | Baseline to Week 52
  After IP administration, the detection of AAV genome was measured using q-PCR.
Evaluation of humoral (anti-AAV9 antibodies) and cellular (IFN-γ activity) immune responses to AAV9 | Baseline to Week 52
  After IP administration, the detection of AAV genome was measured using ELISA
Assessment of AAV9 shedding in biological specimens-urine | Baseline to Week 52
  After IP administration, the detection of AAV genome was measured using q-PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No